CLINICAL TRIAL: NCT02663167
Title: Internet-based Cognitive-behavior Therapy for Children With Obsessive-compulsive Disorder: a Pilot Trial
Brief Title: Internet-based Cognitive-behavior Therapy for Children With Obsessive-compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Serlachius, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPN 2015/470-31
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

ARMS (1):
- Internet-delivered Cognitive-Behavioral Therapy (Experimental)
  Interventions: Behavioral: Internet-delivered Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioral Therapy — The treatment consists of a standard cognitive behavioral therapy for obsessive-compulsive disorder. The treatment is delivered through an Internet platform. The child and his/her parent(s) work through the treatment with regular therapist contact several times per week.

SUMMARY:
The purpose of this study is to evaluate the feasibility and effectiveness of Internet-delivered Cognitive Behavior Therapy (ICBT) for children (7-11 years) with Obsessive-Compulsive Disorder (OCD).

DETAILED DESCRIPTION:
The primary objective of this study is to investigate if Internet-delivered Cognitive Behavior Therapy (ICBT) is a feasible and effective treatment for children (7-11 years) with Obsessive-Compulsive Disorder (OCD). The design of the study is a pilot study with 16 participants. The treatment duration is 12 weeks. The primary outcome measure is the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS). Study participants will be followed up 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-5 diagnosis of OCD
* Total score of ≥16 on the Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS)
* Age between 7-11 years
* Ability to understand Swedish
* Daily access to the Internet
* A parent that can co-participate in the treatment
* Participants on psychotropic medication must had been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* Diagnosed autism spectrum disorder, psychosis, bipolar disorder, severe eating disorder, organic brain disorder, learning disability
* Suicidal ideation
* Not able to understand the basics of the ICBT self-help material
* Have completed a course of CBT for OCD within last 12 months (defined as at least 5 sessions CBT including exposure and response prevention)
* On-going psychological treatment for OCD or another anxiety disorder

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Children´s Yale Brown Compulsive Scale (CY-BOCS) | week 0, week 12, at 3 months follow up
  Change in obsessions and compulsions from baseline to week 12 and at 3 months after treatment has ended

SECONDARY OUTCOMES:
Children's Global Assessment Scale (C-GAS) | week 0, week 12, at 3 months follow up
Clinical Global Impression - Severity (CGI-S) | week 0, week 12, at 3 months follow up
Clinical Global Impression - Improvement (CGI-I) | week 12, at 3 months follow up
Obsessive-Compulsive Inventory - Child Version (OCI-CV) | week 0, week 12, at 3 months follow up and weekly during treatment
Children's Obsessional Compulsive Inventory Revised - Parent version (ChOCI-R-P) | week 0, week 12, at 3 months follow up and weekly during treatment
Family Accommodation Scale - Self Rated (FAS-SR) | week 0, week 12, at 3 months follow up
Euroqol - Youth (EQ-5D-Y) | week 0, week 12, at 3 months follow up
Autism Spectrum Quotient (AQ-10) | week 0
Education, Work and Social Adjustment Scale - child and parent version (EWSAS) | week 0, week 12, at 3 months follow up
Child Depression Inventory - Short version (CDI-S) | week 0, week 12, at 3 months follow up
Mood and Feeling Questionnaire - parent version (MFQ) | week 0, week 12, at 3 months follow up
Qualitative data on treatment credibility | week 3
Qualitative data on treatment satisfaction | week 12
Safety Monitoring Uniform Report Form (SMURF) | week 6, week 12
Internet Intervention Patient Adherence Scale (iiPAS) | week 6, week 12
Patient Exposure/Response prevention Adherence Scale (PEAS) | week 6, week 12

CONTACTS AND LOCATIONS:
Locations (1):
- BUP CPF, Stockholm, Sweden